CLINICAL TRIAL: NCT04299594
Title: Prevalence of Osteoporosis in Sickle Cell Disease
Acronym: DREPAN'OS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0142; 2020-A00490-39 (Other: ID-RDB)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sickle cell disease patients: 150 black patients with sickle cell disease living in France, 20 to 40 years old will be included in this study
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — For each subject recruited, will be collected for the study a questionnaire looking for a history of low energy fracture, and the origins of the patient (or relatives), as well as medical history, lifestyle (alcohol and tobacco consumption), weight and height. This data will be used for the secondary outcomes.

SUMMARY:
Sickle cell disease is the most common single-gene disease in the world. Its prevalence is increasing in France, with patients' life expectancy increasing into developed countries. It mainly affects populations originating from sub-Saharan Africa. Among the chronic bone complications associated with sickle cell disease, osteoporosis has previously been highlighted but remains a poorly known complication in this very particular context. A dedicated evaluation of osteoporosis and associated risk factors in sickle cell disease patients living in France may enable better bone management of these patients in the future, as this problem, specific to their disease, is likely to become more frequent as their life expectancy increases.

This is a prospective interventional and monocentric study whose objective is to describe the prevalence of osteoporosis in black patients with sickle cell disease in France

ELIGIBILITY:
Inclusion Criteria:

* Black-skinned men and women
* Aged 20 to 40 years old
* Sickle cell patients
* Non-opposition to participate in the study

Exclusion Criteria:

* Refusal to participate in the study
* Hemoglobinopathy other than sickle cell disease
* Severe or End Stage Renal Failure
* Long-term corticosteroid therapy (>3 months)
* History of solid cancer or malignant haemopathy
* History of organ transplantation
* Pregnant or breastfeeding woman
* Psychiatric pathology seriously impeding understanding
* Difficulty understanding oral French

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: sickle cell adult patients hospitalized (conventional or day hospitalization) or followed in consultation in internal medicine within the framework of their sickle cell disease at Edouard Herriot Hospital, Lyon, France
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Day 1
  Bone mineral density is measured by systematic bone densitometry at 3 sites: lumbar spine, femoral neck and total hip. These data will be collected in the patient's medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France